CLINICAL TRIAL: NCT04456049
Title: COVID_ENZA Trial: Randomized Open Label Phase II Study to Evaluate the Efficacy of Enzalutamide in High Risk Male Outpatients With COVID-1
Brief Title: Randomized Open Label Phase II Study to Evaluate the Efficacy of Enzalutamide in High Risk Male Outpatients With COVID-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Ricardo Pereira Mestre (Other)
Collaborators: Oncology Institute of Southern Switzerland (Other); Institute of Oncology Research (Unknown); Institute for Research in Biomedicine (Unknown)
Responsible Party: Sponsor-Investigator, Ricardo Pereira Mestre, MD, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID_ENZA
Record Dates: First submitted 2020-07-01; First posted 2020-07-02 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19 | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enzalutamide (Xtandi®) (Experimental): Interventional treatment
  Interventions: Drug: Enzalutamide
- Standard of care (SOC) (Active Comparator): Supportive treatment
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — 40 mg oral tablets once daily for a maximum of 28 days.
  Other Names: XTANDI

SUMMARY:
High risk outpatient adult males with a confirmed SARS-CoV-2 infection will be included in the study.

Patients will be randomized to receive Enzalutamide with standard of care (SOC) or SOC alone. Enzalutamide will be administered daily p.o. from Day 1 to Day 28 or until confirmed negativization of Nasopharyngeal swap (NPS) Polymerase chain reaction (PCR) (2 consecutive negative samples), whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Documented COVID-19 infection (confirmed by NPS positive PCR for SARS-CoV-2) with mild symptoms not requiring hospitalization
* First NPS ≤4 days (96 hours) since onset of symptoms
* Randomization ≤72 hours since first NPS
* Adult Males aged ≥ 50 years
* Indication for outpatient treatment but at high risk for complications, at least 1 risk factor (age ≥ 65 years, hypertension, diabetes, cardiovascular disease, active malignancy, COPD)
* WHO performance status 0-1
* Adequate hematologic values: haemoglobin ≥ 100 g/L, neutrophils ≥ 1.0 x 10(9)/L, platelets ≥ 150 x 10(9)/L.
* Adequate hepatic function: ALT and AST ≤ 2.5 x ULN, bilirubin ≤ 1.5 x ULN (exception if Gilbert's syndrome ≤ 2.5 x ULN)
* Adequate renal function: calculated creatinine clearance ≥ 50 mL/min according to the formula of Cockcroft-Gault
* Patient is able to swallow the trial drugs and to comply with trial requirements
* Patient agrees not to father a child during participation in the trial and for 3 months thereafter

Exclusion Criteria:

* Female sex
* Moderate to severe COVID-19 symptoms requiring hospitalization
* Patients requiring inpatient treatment
* Concurrent antiviral drugs or ongoing interventional clinical trial or any off label drug for COVID-19
* Patients with ongoing prostate cancer treatment
* Clinically significant cardiovascular disease including:

  * Myocardial infarction within 6 months prior to registration,
  * Uncontrolled angina within 3 months prior to registration,
  * Congestive heart failure NYHA class III or VI
  * QTc interval > 480 ms
  * History of clinically significant ventricular arrhythmias (e.g. ventricular tachycardia, ventricular fibrillation, torsades de pointes)
  * History of Mobitz II second or third degree heart block without a permanent pacemaker in place
  * Uncontrolled hypertension as indicated by systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg
  * Deep venous thrombosis or pulmonary embolism within 6 months
  * History of cerebrovascular disease
* Severe concurrent disease, infection or co-morbidity that, in the judgment of the investigator, would make the patient inappropriate for enrolment.
* Known history of HIV, hepatitis B, hepatitis C
* Known history of seizures or any conditions that may predispose to seizure. History of loss of consciousness or ischemic cerebrovascular attack within 12 months prior to registration
* Concurrent anticoagulation with rivaroxaban or warfarin. Concomitant and continuous use of systemic corticosteroids exceeding 10 mg/day of prednisone or a dose equivalent corticosteroid within 14 days before registration.
* Known hypersensitivity to Enzalutamide or hypersensitivity to any of its components
* Any concomitant drugs contraindicated for use with Enzalutamide according to the Swissmedic approved product information
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the trial protocol and follow-up.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of Enzalutamide by decreasing SARS-CoV-2 viral expression | 28 days
  efficacy of Enzalutamide in decreasing the nasopharyngeal swap SARS-CoV-2 viral load until negativization

SECONDARY OUTCOMES:
Tollerability of Enzalutamide by identifying Adverse Events | 28 days
  Evaluation of Enzalutamide tolerability in terms of incidence and severity grade of side effects
Disease progression by unresolved SARS-CoV-2 viral expression after treatment | 28 days
  Efficacy of Enzalutamide in controlling disease progression of SARS-CoV-2 viral load

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Institute of Southern Switzerland (IOSI), Bellinzona, Switzerland